CLINICAL TRIAL: NCT00318552
Title: Pharmacoeconomic Analysis of First Line Meropenem Versus Standard Antibiotic Treatment in Seriously Infected Secondary Nosocomial Sepsis Syndrome Patients. An Open, Randomized Multi-center Study.
Brief Title: Pharmacoeconomic Analysis of First Line Meropenem Versus Standard Antibiotic Treatment in Seriously Infected Secondary Nosocomial Sepsis Syndrome Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3591/9014; D9211C09014 (Other: AZ IMPACT)
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Sepsis
Keywords: Antibiotic Therapy; sepsis treatment; Meropenem
MeSH Terms: conditions — Sepsis | interventions — Meropenem

INTERVENTIONS:
Drug: Meropenem

SUMMARY:
This study will directly compare meropenem with standard first line antibiotic therapies in subjects entering an ICU with secondary nosocomial sepsis, or who contract sepsis while resident in an ICU.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥ 18, requiring intensive care treatment related to secondary nosocomial sepsis, who require potent broad spectrum intravenous antibiotic therapy.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2002-01; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Number of days from randomization to recovery from sepsis among those patients who survived the trial period
Endpoint considered in conjunction with observed mortality rates to determine whether any reduction in time to recovery from sepsis

SECONDARY OUTCOMES:
Number of days from randomization to ready to discharge from the ICU
Number of days from randomization until patient is discharged from the ICU
Number of days on first line antibiotic therapy
Number of days from randomization until patient is discharged from hospital
Proportion of patients who achieve clinical cure from sepsis following first line antibiotic therapy
Proportion of all patients who are ready to discharge from the ICU following antibiotic therapy
Mortality rate due to "all causes" in the meropenem group and the standard antibiotic therapy group
Mortality rate due to infection in the meropenem group and the standard antibiotic therapy group
Health Economics-Resource utilization for main treatment and diagnostic procedures, tools and materials

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca CRR Central and Eastern Europe, Hungary Medical Director, MD, Study Director — AstraZeneca
Locations (12):
- Hungary (12):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Eger
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Siófok
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Veszprém